CLINICAL TRIAL: NCT00124384
Title: Phase 4 Study of the Effects of Modafinil on Waking Function and on Sleep in Individuals With Primary Insomnia
Brief Title: The Effects of Modafinil on Waking Function and on Sleep in Individuals With Primary Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Michael L. Perlis, PhD., University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1538a/6029/IN/US; RSRB # 10306
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Primary Insomnia
Keywords: primary insomnia, stimulants, cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: CBT-I
Drug: modafinil

SUMMARY:
This study examines how treatment with the drug modafinil, by itself or in combination with cognitive behavioral treatment for insomnia (CBT-I), may improve daytime functioning and/or diminish the severity of insomnia.

DETAILED DESCRIPTION:
Our primary goal is to undertake a 2nd study evaluating whether Modafinil, alone or in combination with behavioral treatment for insomnia, will improve subjects' sleep continuity and/or self report daytime function.

METHODS AND PROCEDURES

Schedule for Procedures.

Screening interview Sleep over night in our lab for one night 8 weeks of either behavioral or psychological therapy for insomnia 3 month post therapy follow up (two weeks of sleep diaries and one lab visit)

40 patients aged 25-80 with insomnia. All subjects will have a stable sleep/wake schedule with a preferred sleep phase between 10:00 PM and 8:00 AM. The age range is restricted to 1) minimize circadian rhythm influences on the diagnoses of Psychophysiological insomnia, 2) to increase our ability to recruit medically healthy sample, and 3) increase sample homogeneity.

All subjects will meet diagnostic criteria for Psychophysiological Insomnia according to the International Classification of Sleep Disorders (ICSD). Criteria are: the complaint of insomnia and impaired daytime function; an indication of learned sleep-preventing associations and somatized tension; active help seeking. The complaint of disturbed sleep will have one or more of the following characteristics: >30 minutes to fall asleep and/or >2 awakenings per night of >15 minutes duration and/or wake after sleep onset time of > 30 minutes, problem frequency >4 nights/ week, and problem duration >6 months. In addition, all subjects will complain of fatigue and/or sleepiness at intake.

Treatment.

Regardless of group assignment, all subjects will 1) wear an actiwatch, 2) be seen on an individual basis for 8 weeks. Session length will be held constant and all patients will be seen by the same therapist (Wilfred Pigeon, PhD). Backup support will be provided by the Principal Investigator (Michael Perlis, PhD) or by the Clinic's Nurse Practitioner (Carla Jungquist, MSN) and 3) complete daily sleep diaries for duration of the study (from study intake until study end [8 weeks]).

ELIGIBILITY:
Inclusion Criteria:

* 40 patients aged 25 with insomnia, will be recruited over a 3-6 month interval.
* All subjects will have a stable sleep/wake schedule with a preferred sleep phase between 10:00 PM and 8:00 AM.
* Must live in the Greater Rochester NY area
* All subjects will meet diagnostic criteria for Psychophysiological Insomnia according to the International Classification of Sleep Disorders (ICSD). Criteria are: the complaint of insomnia and impaired daytime function; an indication of learned sleep-preventing associations and somatized tension; active help seeking. The complaint of disturbed sleep will have one or more of the following characteristics: >30 minutes to fall asleep and/or >2 awakenings per night of >15 minutes duration and/or wake after sleep onset time of > 30 minutes, problem frequency >4 nights/ week, and problem duration >6 months. In addition, all subjects will complain of fatigue and/or sleepiness at intake.

Exclusion Criteria:

* As above

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in sleep latency, wake after sleep onset, sleep efficiency; efficacy of modafinil and the combination of modafinil and CBT-I on previously mentioned outcome measures

SECONDARY OUTCOMES:
Long term (3 months) effects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perlis, PhD, Principal Investigator — University of Rochester Sleep Research Lab
Locations (1):
- University of Rochester Sleep and Neurophysiology Research Lab, Rochester, New York, United States

REFERENCES:
- [Background] Perlis ML, Smith MT, Orff H, Enright T, Nowakowski S, Jungquist C, Plotkin K. The effects of modafinil and cognitive behavior therapy on sleep continuity in patients with primary insomnia. Sleep. 2004 Jun 15;27(4):715-25. doi: 10.1093/sleep/27.4.715. PMID 15283007